CLINICAL TRIAL: NCT05083715
Title: The Impact of the Head Position on the Occlusion of Implant-supported Fixed Restorations vs. Natural Dentition - a Cross-sectional Analysis
Brief Title: The Impact of the Head Position on the Occlusion of Implant-supported Fixed Restorations
Acronym: TIOTHPOTO
Status: Completed | Type: Observational
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Ana Todorovic, Senior Lecturer, University of Belgrade
Other Study IDs: Univerzitet Beograd
Record Dates: First submitted 2021-10-05; First posted 2021-10-19 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Dental Occlusion
Keywords: dental occlusion; head posture; fixed dental restorations; dental implants; implant occlusion; computerized occlusal analysis
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The development of a implantology leads to an increasing use of implants in the treatment of care for the loss of one or more teeth. The question is whether the existing guidelines, originally formulated for the occlusion of natural dentition and conventional prosthetic treatment can be applied to the implant prosthodonticsDue to initial differences in the vertical mobility of teeth and dental implants, present in the same dental arch, although the model of occlusion is ideal, undesirable premature occlusal contacts on the fixed dental restorations on implants may be present.

Objective: To evaluate the effect of different head positions on dental occlusion of the natural teeth and fixed dental restorations on implants.

Methods: Volunteers with complete dentition would be included in this study as the Control Group. The Study Group would include subjects with fixed dental restorations on implants in the transcanine region. A T Scan III System will be used for occlusal analysis.

ELIGIBILITY:
Inclusion Criteria:

For the Test Group

* patients with implant-supported fixed restorations in at least one quadrant of the posterior region (pre-molar and molar) of both jaws at least for 1 year
* patients with Angle Class I in MIP
* patients who did not have orthodontic treatment

For the Control group, the inclusion criteria were:

- patients with completely dentate arches (not considering third molars) with a maximum of 4 tooth-supported restorations per dental arch).

Exclusion Criteria:

* patients with bruxism, detrimental habits, and mandibular parafunctional activities
* patients with signs of temporomandibular dysfunction, trismus, or illness of the cervical spine
* patients with a history indicating problems with alcohol or drugs or receiving any psychiatric treatment.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who refered to the Clinic for Prosthodontics due to the lack of one or more teeth that need to be replaced with dental implants and healthy completely dentate volunteers.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Changes in occlusal contacts distribution in 3 different head positions | Baseline-1 year
  Computerized occlusal analysis
Changes in relative forces strength in 3 different head positions | Baseline-1 year
  Computerized occlusal analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ana R Todorovic, DDS,PhD, Principal Investigator — Clinic for Prosthodontics, University of Belgrade Serbia
Locations (1):
- Clinic for Prosthodontics, University of Belgrade Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldstein G, Goodacre C, Taylor T. Occlusal Schemes for Implant Restorations: Best Evidence Consensus Statement. J Prosthodont. 2021 Apr;30(S1):84-90. doi: 10.1111/jopr.13319. PMID 33783094
- [Background] Sadowsky SJ. Occlusal overload with dental implants: a review. Int J Implant Dent. 2019 Jul 23;5(1):29. doi: 10.1186/s40729-019-0180-8. PMID 31332553
- [Background] Afrashtehfar KI, Qadeer S. Computerized occlusal analysis as an alternative occlusal indicator. Cranio. 2016 Jan;34(1):52-7. doi: 10.1179/2151090314Y.0000000024. Epub 2014 Oct 16. PMID 25323220
- [Background] Chapman RJ, Maness WL, Osorio J. Occlusal contact variation with changes in head position. Int J Prosthodont. 1991 Jul-Aug;4(4):377-81. PMID 1811633